CLINICAL TRIAL: NCT02247037
Title: Patient-derived Xenograft (PDX) Modeling of Treatment Response for Triple Negative Breast Cancer
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Champions Oncology (Industry)
Responsible Party: Principal Investigator, Hanna Irie, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 14-0686
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple Negative Breast Cancer; Patient Derived Xenograft; Neoadjuvant Chemotherapy; Therapeutic Resistance
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Core Biopsy Specimen, Surgical Specimen
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Triple Negative Breast Cancers: All women eligible for this protocol will fall into this group. These women will have histologically confirmed triple negative breast cancer and be eligible for neoadjuvant chemotherapy or have evidence of metastatic disease.
  Interventions: Other: Chemotherapy

INTERVENTIONS:
Other: Chemotherapy — Patients are treated with neoadjuvant chemotherapy as according to the standard of care guidelines. Patients with metastatic disease are treated according to standard of care guidelines.

SUMMARY:
This study will determine if patient-derived tumor xenograft (PDX) mouse models can serve as a reliable model for treatment response for individual patients with triple negative breast cancer. The collection of patient tumor tissue will also provide insight into the mechanisms of therapeutic resistance for those individuals. Ultimately, this study will enhance our understanding of the genomic basis for treatment response for triple negative cancer on an individual basis, while having the potential to suggest new therapeutic options for high-risk triple negative breast cancer patients with residual disease post neoadjuvant.

DETAILED DESCRIPTION:
Triple negative breast cancer (TNBC) represents an aggressive, genomically heterogeneous, subtype of breast cancer with limited therapeutic options. Many patients with TNBC receive standard neoadjuvant chemotherapy (NAC) pre-operatively; response is directly correlated with long-term outcome. Patients with residual disease after NAC are at higher risk for recurrent or metastatic disease, but additional adjuvant therapies are not currently part of standard care. Personalized treatment for patients with TNBC requires an improved understanding of the genomic landscape of individual TN breast tumors, as well as improved predictive models of response to specific therapeutic agents. This pilot study will determine if patient-derived tumor xenograft (PDX) mouse models can serve as a reliable model for treatment response for individual patients with TNBC. The tumor tissue collected (paired pre-and post NAC) will also provide insight into mechanisms of therapeutic resistance for individual patients. This study will enhance our understanding of the genomic basis for treatment response for TNBC on an individual patient basis, and lead to potential new therapeutic options for high-risk TNBC patients with post-NAC residual disease.

Objectives:

1. To collect and bank tissue specimens from patients with operable triple negative breast cancer at: a) at time of diagnosis, prior to the start of neoadjuvant therapy and b) at time of definitive surgery, after the completion of neoadjuvant therapy.
2. To collect and bank tissue specimen for patients with advanced metastatic triple negative disease prior to start of any line therapy for metastatic disease.
3. To create patient-derived xenograft (PDX) mouse models utilizing specimens collected pre- and post- neoadjuvant treatment
4. To determine if response of PDX tumors to cytotoxic agents in the Champions Oncology Tumor GraftTM (COTG) assay correlates with responses observed in patients.
5. To perform genomic analyses of patient tumor specimens collected pre- and post neoadjuvant treatment to study mechanisms of drug resistance

ELIGIBILITY:
Inclusion Criteria:

* a histological diagnosis of invasive triple negative breast cancer determined by standard immunohistochemical analysis.
* must be candidates for neoadjuvant chemotherapy according to standard of care guidelines or have evidence of metastatic disease.
* must agree to a biopsy for research purposes at time of diagnosis and to undergo surgery at the hospitals of the Mount Sinai Health System.

Patients with the following MAY be eligible:

- a histological diagnosis of ER and/or PR positive breast cancer with an overall receptor expression ≤ 30% breast cancer determined by standard immunohistochemical analysis

Exclusion Criteria:

* concurrent disease or condition that would make the patient inappropriate for study participation,
* any serious medical or psychiatric disorder that would interfere with the subject's safety, or inability to provide informed consent.
* vulnerable populations will not be included.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Triple Negative Breast Cancer that are eligible for neoadjuvant chemotherapy or have evidence of metastatic disease will be pursued for this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2014-07; Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Patient Tumor Response | Day 1
  Tumor response in patients will be categorized as: Progressive Disease, Static Response, Partial Response, Complete Response

SECONDARY OUTCOMES:
Model Tumor Response | Day 1
  Tumor response in models will be categorized as: Progressive Disease, Static Response, Partial Response, Complete Response

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Yoko Irie, MD, PhD, Principal Investigator — Dubin Breast Center of The Tisch Cancer Institute at Mount Sinai; Elisa Port, MD, Principal Investigator — Dubin Breast Center of The Tisch Cancer Institute at Mount Sinai
Locations (1):
- Dubin Breast Center of The Tisch Cancer Institute at Mount Sinai, New York, New York, United States